CLINICAL TRIAL: NCT01103453
Title: Change in Executive Functions and in Instrumental Activities of Daily Living as a Result of Intervention by Virtual Supermarket Environment Among People With Mild Cognitive Impairment.
Brief Title: Change in Executive Function and IADL Using a Virtual Supermarket Environment Among People With MCI
Acronym: EF-VAPS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Dr Gary Sinoff, Director Cognitive Clinic, Carmel Medical Center, Haifa, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMC090105CTIL
Record Dates: First submitted 2010-04-07; First posted 2010-04-14 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Mild Cognitive Impairment; Lack of Physical Activity
Keywords: MCI; Executive Function; ADL; Virtual Supermarket
MeSH Terms: conditions — Cognitive Dysfunction; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Group (Experimental): Study group are persons diagnosed as suffering from Mild Cognitive Impairment will undergo a series of 9 sessions on a computer program of a virtual supermarket to improve their Executive and IADL functions.
  Interventions: Behavioral: Virtual Action Planning Supermarket (VAP-S) Software

INTERVENTIONS:
Behavioral: Virtual Action Planning Supermarket (VAP-S) Software — The VAP-S simulates a supermarket with multiple aisles displaying items. Several obstacles are designed to hinder the progression of the shopper along the aisles. In addition, virtual humans populate the supermarket. The VAP-S is designed so that the user enters the supermarket behind the cart and navigates within the supermarket via the keyboard keys. He is thus able to experience the environment personally without any intermediate. The task is to purchase 7 items from a list, proceed to the cashier and pay for them.
  We propose 9 sessions of 45 minutes. The results will be analyzed to develop goals for intervention, together with the client to study his awareness of his performance of IADL and Executive functions and to enhance his motivation to participate in the intervention.
  Other Names: VAP-S Virtual Action Planning - Supermarket; Virtools Development - Interactive 3D Development Tool; Discreet 3D Studio Max4 Graphics

SUMMARY:
The aim of the study is to investigate the feasibility of using a virtual supermarket as an intervention tool for overcoming deficits in executive function as well as enhancing IADL performance among persons with Mild Cognitive Impairment. The working hypotheses are that there will be improvement in executive functions, and the improvement in the executive functions will result in better performance in Instrumental Activities of Daily Living, both generally and especially in shopping task

DETAILED DESCRIPTION:
Scientific and clinical research in the area of Alzheimer's disease (AD) during the last years have shifted their focus to earlier diagnosis and especially to the transitional phase between normal aging and dementia, named Mild Cognitive Impairment (MCI).Lately, the concept of MCI has been expanded to address observed clinical heterogeneity, and subtypes were recognized: amnestic (including memory impairment) and non-amnestic (including impairment in other non-memory cognitive domains), with the later including deficits in executive functioning Executive functions (EF) are defined as higher order functions that are needed for completing complex or non-routine tasks. Deficits in EF refer to a collection of deficits in attention, planning, problem-solving, multitasking, monitoring and behavioral control and persons who suffer from impairments in EF typically have difficulty in initiating or suspending activities, show impaired mental flexibility, as well as increased distractibility and have difficulty in learning novel tasks despite apparently intact cognitive abilities.

Lately, an increasing amount of studies suggest that persons with MCI might have deficits in EF, moreover, persons presenting a combination of executive deficits and memory deficits were found to be a high risk group for conversion to AD.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+
* Diagnosed as suffering from MCI
* No impaired judgement
* Verbal and written proficiency in Hebrew
* Normal or corrected-to-normal vision and hearing ability
* Independent in ADL function
* Lives in the community
* Able to perform task of shopping.

Exclusion Criteria:

* Suffering from other coexistent neurological diseases (e.g. stroke, muscular dystrophy)
* Has acute arthritis
* Poorly controlled hypothyroidism
* Suffering from physical or sensory limitations, as by self-report or noted by the investigator, that may limit the use of a computer's mouse
* No skills in performing shopping task
* Defined as suffering from depression as determined by the rating scale for depression
* Diagnosed as suffering from dementia as defined by Diagnostic and Statistical Manual of Mental Disorders criteria (DSM-IV)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in executive functions by means of comparison to the results on the NexAde® computerized test. | 1 month after intervention
  The NexAde® is a computerized assessment test for deficits in cognition and executive function. The test consists of several neuropsychological tests used in clinical practice and research and the domains being assessed are attention, memory, visuomotor learning, spatial memory, executive function and mental flexibility. The test has been adapted for older adults who are not familiar with computers and was found to be reliable and valid.

SECONDARY OUTCOMES:
Improved performance in IADL, both generally and especially in shopping task. | 1 month after intervention
  IADL will be examined by means of results on the MET (Multiple Errands Test) and Lawton and Brody's IADL instruments. The MET assesses executive function while performing an everyday activity by observation. It consists of three main tasks in shopping: purchase six items, find out four different pieces of information and meet the examiner at a specific time at a predetermined location. Lawton & Brawdy's IADL instrument evaluates the subject's capacity to perform eight different IADL tasks such as cooking, the use of transportation and shopping.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Sinoff, MD, PhD, Principal Investigator — Carmel Medical center, Haifa, Israel
Locations (1):
- Cognitive Clinic, Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Belleville S. Cognitive training for persons with mild cognitive impairment. Int Psychogeriatr. 2008 Feb;20(1):57-66. doi: 10.1017/S104161020700631X. Epub 2007 Oct 25. PMID 17958927
- [Background] Sgaramella TM, Borgo F, Mondini S, Pasini M, Toso V, Semenza C. Executive deficits appearing in the initial stage of Alzheimer's disease. Brain Cogn. 2001 Jun-Jul;46(1-2):264-8. doi: 10.1016/s0278-2626(01)80080-4. PMID 11527345
- [Background] Josman N, Schenirderman AE, Klinger E, Shevil E. Using virtual reality to evaluate executive functioning among persons with schizophrenia: a validity study. Schizophr Res. 2009 Dec;115(2-3):270-7. doi: 10.1016/j.schres.2009.09.015. Epub 2009 Oct 22. PMID 19850451
- [Background] Werner P, Rabinowitz S, Klinger E, Korczyn AD, Josman N. Use of the virtual action planning supermarket for the diagnosis of mild cognitive impairment: a preliminary study. Dement Geriatr Cogn Disord. 2009;27(4):301-9. doi: 10.1159/000204915. Epub 2009 Mar 2. PMID 19252401